CLINICAL TRIAL: NCT05137262
Title: Durvalumab and Standard Chemotherapy for the Treatment of Lymph Node Positive Bladder Cancer
Brief Title: A Phase II Multicenter Study of Chemotherapy Versus Chemotherapy Plus Durvalumab (MEDI 4736) in Patients With Lymph Node Positive Urothelial Carcinoma of the Bladder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1091; NCI-2021-12884 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Urothelial Carcinoma; Bladder Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — Abiraterone Acetate; durvalumab; Methotrexate; Vinblastine; Doxorubicin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Standard of Care with dose-dense MVAC (Experimental): The patient will receive treatment every 14 days for up to 6 cycles in the neoadjuvant setting.
  Interventions: Other: Abiraterone acetate; Drug: Durvalumab; Drug: Methotrexate; Drug: Vinblastine; Drug: Doxorubicin Hydrochloride; Drug: Cisplatin
- Arm B: Intervention with dose-dense MVAC plus Durvalumab (Experimental): Durvalumab will be administered one week prior to the initial cycle of dose-dense MVAC and then with each additional cycle of dose-dense MVAC on Arm B
  Interventions: Other: Abiraterone acetate; Drug: Durvalumab; Drug: Methotrexate; Drug: Vinblastine; Drug: Doxorubicin Hydrochloride; Drug: Cisplatin

INTERVENTIONS:
Other: Abiraterone acetate — Given by IV
  Other Names: Zytiga™
Drug: Durvalumab — Given by IV
  Other Names: MEDI4736
Drug: Methotrexate — Given by IV
Drug: Vinblastine — Given by IV
  Other Names: Velban
Drug: Doxorubicin Hydrochloride — Given by IV
  Other Names: Adriamycin RDF™; Adriamycin PFS®; Adriamycin®; Rubex®
Drug: Cisplatin — Given by IV
  Other Names: Platinol®-AQ; Platinol®; CDDP

SUMMARY:
This is a phase II randomized study of standard of care (SOC) neo-adjuvant cisplatin chemotherapy (NAC) versus NAC plus durvalumab in patients with either clinical or pathologic intra-pelvic node-positive urothelial carcinoma of the bladder. Patients with cTanyN1-3M0 via American Joint Committee on Cancer (AJCC) 8th edition staging30 will be considered tor enrollment in this trial. We plan to enroll 60 patients. Patients will be randomized 2:1 to the intervention arm with durvalumab plus NAC vs SOC NAC. In patients randomized to receive, durvalumab will be continued as maintenance every 4 weeks until either relapse or 1 year, whichever event occurs first.

Tissue collection will occur as a biopsy prior to initiation of neo-adjuvant therapy via both transurethral biopsy of bladder and lymph node biopsy. Tissue will again be collected at the time of radical cystectomy or, in patients who are no longer surgical candidates, in the form of biopsy as standard of care. Blood and urine will be collected at baseline, week 2, week 6, week 16, and at the 6 week-post surgery visit for analysis of correlative studies.

DETAILED DESCRIPTION:
Primary Objective:

• To estimate the difference in pathologic complete response rate as defined as no evidence of disease (ypT0N0) or carcinoma in situ within the bladder only (ypTcisN0) in patients after administration of the combination of dose-dense MVAC and durvalumab versus dose-dense MVAC alone.

Secondary Objectives:

* To estimate the difference in the rate of patients eligible for surgical consolidation within 90 days of completion of pre-surgical treatment.
* To estimate the difference in the proportion of patients with relapse free survival at 12 and 36 months following surgery in each treatment arm.
* To estimate the difference in overall survival for both arms on study.
* To measure lymph node response with those with measurable disease via RECIST v1.1 criteria at baseline, week 6, and week 12 on study.
* To evaluate the toxicity of the combination of dose-dense MVAC chemotherapy and durvalumab.

Correlative Objectives:

• Exploratory biomarkers to study the correlation between immunological and molecular changes in tumor tissues and peripheral blood with pathologic complete response, time until relapse and rate of adverse events, with a specific emphasis upon comparison of tissue samples in patients exposed to combination dose-dense MVAC and durvalumab versus dose-dense MVAC alone

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological diagnosis of urothelial carcinoma of the bladder and must meet criteria for stage cTanyN1-3M0 disease via AJCC 8th edition staging criteria30
* Patients must provide tissue by agreeing to transurethethral biopsy of the bladder and the lymph node prior to initiating treatment. If patient is unable or unwilling to undergo biopsy at screening and tissue is available, patient may be eligibile per PI discretion.
* Patients must be ≥18 years of age.
* Patients must have pelvic lymph node amenable for biopsy as assessed by treating MD and interventional radiologist.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must have body weight >30 kg.
* Left ventricular ejection fraction ≥ 50%.
* Adequate organ function as defined below:

  * Hematological i. Absolute neutrophil count (ANC) ≥ 1,500/mcL. ii. Platelets ≥100,000 / mcL. iii. Hemoglobin ≥9 g/dL
  * Renal iv. Creatinine clearance > 50 ml/min as calculated by the Cockgroft Gault formula as:

    1. CLCR = {[(140-age) × weight)]/(72 x SCR) × 0.85 (if female), where CLCR (creatinine clearance) is measured in mL/min, age is expressed in years, weight in kilograms (kg), and SCR (serum creatinine) in mg/dL.
  * Hepatic v. Serum total bilirubin ≤1.5xULN OR Direct bilirubin ≤ULN for subjects with total bilirubin levels >1.5xULN. vi. AST and ALT ≤2.5xULN OR ≤5xULN for subjects with liver metastases.
  * Coagulation vii. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5xULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants. viii. Activated Partial Thromboplastin Time (aPTT) ≤1.5xULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
* Women of child-bearing potential MUST have a negative serum or urine HCG test unless prior tubal ligation (>/= 1 year before screening), total hysterectomy or menopause (defined as 12 consecutive months of amenorrhea). Patients should not become pregnant or breastfeed while on this study. Sexually active patients must agree to use dual contraception for the duration of study participation and for 90 days after receipt of last drug on active treatment.
* Ability to understand and willingness to sign informed consent from prior to initiation of the study and any study procedures.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Has metastatic disease to lymph nodes outside of the pelvis or to visceral sites as seen on imaging.
* CTCAE v5.0 Grade ≥ 2 neuropathy.
* CTCAE v5.0 Grade ≥ 2 hearing loss.
* New York Heart Association (NYHA) Class III or IV heart failure defined as:

  * Class III heart failure is defined as: patients with cardiac disease resulting in marked limitation of physical activity and/or less than ordinary activity causes fatigue. Patients are comfortable only at rest.
  * Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases
* Known active Hepatitis B, Hepatitis C infection (HCV-DNA positive), or HIV infection.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of study drug, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Systemic steroid administration required to manage toxicities arising from chemotherapy and/or immunotherapy delivered as part of the therapy on trial is allowed.
* Prior exposure to any anti-PD-1 or anti-PD-L1 (including durvalumab) antibody.
* Active or prior documented autoimmune disease within the past 2 years. NOTE: Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* History of primary immunodeficiency.
* History of allogeneic organ transplant.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note:

Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.

* Active infection requiring intravenous (IV) antibiotics or other uncontrolled intercurrent illness requiring hospitalization. Minor infections, e.g. periodontal infection or urinary tract infection (UTI), which may be treated with short-term oral antibiotics are allowed.
* Active infection of tuberculosis, as determined by clinical signs and symptoms.
* Inability to comply with the study and follow-up procedures.
* History of CVA, myocardial infarction or unstable angina within the previous 6 months before starting therapy.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* Has a known additional malignancy that is progressing or requires active treatment.

Exceptions include basal cell carcinoma of the skin, organ confined adenocarcinoma of the prostate, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. Patients may not have received systemic cytotoxic chemotherapy within 1 year of study entry.

* History of exposure to immunotherapy for previous malignancy.
* Intra-vesicular therapy within 4 weeks of study entry or those who have not recovered from adverse effects of such agents administered more than 4 weeks earlier.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to methotrexate, vinblastine, doxorubicin, cisplatin, durvalumab, or any other agents used in the study.
* Pregnant female patients; breastfeeding female patients; and female or male patients of childbearing potential who are unwilling or unable to use 2 methods of contraception for at least 90 days after the last dose of study drugs. Highly effective methods of contraception are those that alone or in combination, result in a failure rate of less than 1% per year when used consistently and correctly. These methods include:
* Established use of oral, inserted, or injected or implanted hormonal methods of contraception are allowed provided the patient remains on the same treatment throughout the entire study and has been using that hormonal contraceptive for an adequate period of time to ensure effectiveness.
* Correctly placed copper containing intrauterine device (IUD).
* Male condom or female condom used with spermicide (i.e. foam, gel, film, cream or suppository).
* Male sterilization with appropriately confirmed absence of sperm in the post vasectomy ejaculate.
* Bilateral tubal ligation or bilateral oophorectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
To estimate the difference in the pathologic complete response rate. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Campbell, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Indiana University, Bloomington, Indiana
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org